CLINICAL TRIAL: NCT06310356
Title: Continuous Glucose Monitoring for Women with Gestational Diabetes: a Randomized Controlled Trial
Brief Title: Continuous Glucose Monitoring for Women with Gestational Diabetes
Acronym: CORDELIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); General Hospital Groeninge (Other); Onze Lieve Vrouw Hospital (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Vitaz (Other); Centre Hospitalier Universitaire de Liege (Other); Erasme University Hospital (Other); Université Catholique de Louvain (Other); University Hospital, Ghent (Other); AZ Sint-Lucas Gent (Other); AZ Sint-Lucas Brugge (Other); AZ St Maarten Mechelen (Unknown); Imelda Hospital, Bonheiden (Other); AZ Oostende (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORDELIA
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; continuous glucose monitoring; early gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous glucose monitoring (Experimental): continuous use of realtime-continuous glucose monitoring with Freestyle Libre 3
  Interventions: Device: Freestyle Libre 3
- self monitoring of blood glucose with glucometer (Active Comparator): self monitoring of blood glucose with glucometer, at least 2 days per week if treated with lifestyle and daily if additional treatment with insulin is started
  Interventions: Device: Glucometer

INTERVENTIONS:
Device: Freestyle Libre 3 — CGM
  Arms: continuous glucose monitoring
Device: Glucometer — SMBG
  Arms: self monitoring of blood glucose with glucometer

SUMMARY:
There are a few ongoing large randomized controlled trials (RCT's) on continuous glucose monitoring (CGM) in women with gestational diabetes (GDM) powered for pregnancy outcomes. However, none of these studies included women diagnosed with early GDM. The CORDELIA trial is a Belgian open-label multi-centric RCT with 14 centers in women with GDM (including both early and late GDM). Women will be randomized 1/1 to either treatment with CGM (intervention group, Freestyle Libre 3) or continue with self-monitoring of blood glucose (SMBG) with glucometer in line with normal routine (control arm). The study ends at the postpartum oral glucose tolerance test (OGTT 6-24 weeks postpartum) to screen for glucose intolerance.

DETAILED DESCRIPTION:
At diagnosis of GDM, women will receive education on the management of GDM with lifestyle and need to monitor glucose with SMBG. Within one week of GDM diagnosis, all participants will be asked to use a blinded CGM (Freestyle Libre Pro IQ,) during a run-phase. Women randomized to the control arm, will be asked to intermittently wear a blinded CGM sensor (Freestyle Libre Pro IQ) during 14 days at least two time points in pregnancy (at 31.0-33.6 weeks and between 36.0-38.6 weeks). For women diagnosed with early GDM (<20 weeks), blinded CGM will be needed 3 times in pregnancy with a first time at 20.0-23.9 weeks. Women randomized to the intervention arm will be recommended tu use the rt-CGM (Freestyle Libre 3) till the delivery. In line with normal routine, a 75g OGTT will be performed between 6-24 weeks postpartum to screen for glucose intolerance. Participants will be asked to also wear a blinded CGM (Freestyle Libre Pro IQ) at this last study visit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the Informed Consent Form (ICF)
* Singleton pregnancy
* Diagnosed with gestational diabetes before 29.6 weeks of pregnancy
* Needs to be able to understand and speak Dutch, French or English.
* Have email access

Exclusion Criteria:

* Patient has a history of type 2 or type 1 diabetes, or presence of auto-immune antibodies for type 1 diabetes
* A physical or psychological disease likely to interfere with the conduct of the study (based on the evaluation by the treating physician).
* Use of medication with significant impact on glycemia (such as high dose glucocorticoids and diabetes medication such as metformin)
* Participation in an interventional Trial with an investigational medicinal product or device
* Multiple pregnancy
* History of bariatric surgery
* Known allergy to the adhesives used with the continuous glucose monitoring

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 386 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
a composite of pregnancy outcomes | at delivery
  Hence, the primary outcome is a binary variable, taking the value 1 if at least one of the adverse pregnancy outcomes occurs, or zero otherwise:preterm delivery <37 weeks, large-for-gestational age infant, neonatal hypoglycaemia, (requiring intravenous dextrose), NICU admission (>24h), respiratory distress (at least 4 hours of respiratory support with supplemental oxygen, CPAP, or intermittent positive-pressure ventilation during the first 24 hours after delivery), stillbirth or neonatal death, phototherapy for jaundice, birth trauma and shoulder dystocia

SECONDARY OUTCOMES:
time in glucose range overnight between 70-95mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 00 till 6am between 70-95mg/dl
time in glucose range during the day between 70-95mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 06 am til 00 between 70-95mg/dl
time in glucose range overnight between 63-140mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks of gestation
  time in range from 00 till 6am between 63-140mg/dl
time in glucoserange during the day between 63-140mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 06 am til 00 between 63-140mg/dl
time in glucose range during the day between 54-95mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 06 am til 00 between 54-95mg/dl
time in glucose range overnight between 54-95mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 00 till 6am between 54-95mg/dl
time in glucose range overnight between 63-120mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 00 till 6am between 63-120mg/dl
time in glucose range during the day between 63-120mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 06 am til 00 between 63-120mg/dl
hypoglycemia <54mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time below 54mg/dl
hypoglycemia <50mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time below 50mg/dl
hypoglycemia <63mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time below 63mg/dl
hypoglycemia <70mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time below 70mg/dl
standard deviation | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  glycemic variability measured by standard deviation (SD)
Coefficient of Variance | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  glycemic variability measured by coefficient of variance (CV)
mean amplitude of glycemic excursions | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  glycemic variability measured by mean amplitude of glycemic excursions (MAGE)
glucose time overnight >100mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time in range from 00 till 6am >100mg/dl
glucose postprandial time >120mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  postprandial time >120mg/dl 2hours after the meal
glucose postprandial time >140mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  postprandial time >140mg/dl 1hour after the meal
glucose time >180mg/dl | during 2 weeks between 20.0-23.6 weeks, 31.0-33.6 weeks, and 36.0-38.6 weeks
  time >180mg/dl
mean HbA1c | between 20.0-23.6 weeks, 31.0-33.6 weeks, 36.0-38.6 weeks and 6-24 weeks postpartum
  glycated Hb
Glucose management indicator | between 20.0-23.6 weeks, 31.0-33.6 weeks, 36.0-38.6 weeks and 6-24 weeks postpartum
  Glucose management indicator, GMI
timing of start insulin treatment | from GDM diagnosis till delivery
  gestational age at start insulin treatment
mean insulin dose | from GDM diagnosis till delivery
  dose of short and/or long)actinbg insulin
mean gestational weight gain | at delivery
  weight gain in pregnancy
rate of postpartum hemorrhage | at delivery
  hemorrhage with delivery
rate of macrosomia | at delivery
  birth weight >4Kg
rate of baby >4.5Kg | at delivery
  birth weight >4.5Kg
rate of Small-for-gestational age infant | at delivery
  birth weight <10Th percentile
rate of cesarean section | at delivery
  total (planned and emergency) number of cesarean sections
rate of instrumental delivery | at delivery
  delivery with forceps or vacuum
rate of perineal inury | at delivery
  3dr or 4th degree perineal laceration
rate of labor inductions | at delivery
  induction of labor
rate of preeclamspia | at delivery
  [≥20 weeks of gestation: new onset of hypertension and proteinuria or the new onset of hypertension and significant end-organ dysfunction with or without proteinuria (dipstick ≥ 2+, ≥0.3 g protein/24 hours or ≥30 mg/dL protein in spot urine or spot urine protein / creatinine ratio ≥30 mg protein/mmol creatinine
rate of gestational hypertension | at delivery
  ≥20 weeks of gestation: blood pressure ≥140/90mmHg
rate of fetal malformation | at delivery
  congenital malformation
rate of miscarriage | at delivery
  fetal loss <20 weeks gestation
rate of polycythemia | at delivery
  increased hematocrite accoridng to local practice
rate of neonatal hypoglycemia | at delivery
  bypoglycemia at birth <40mg/dl
Treatment satisfaction | between 31.0-33.6 weeks, 36.0-38.6 weeks and 6-24 weeks postpartum
  diabetes treatment satisfaction questionnaire score, the higher the score the more satisfied, max. score of 48
Quality of life based on Short Form (SF-36) score | baseline, between 36.0-38.6 weeks and 6-24 weeks postpartum
  Short Form (SF-36) score, the higher the score the higher the Quality of life with a max score of 100
dietary intake | baseline, between 36.0-38.6 weeks and 6-24 weeks postpartum
  Frequyency Food Questionnaire
Physical activity | baseline, between 36.0-38.6 weeks and 6-24 weeks postpartum
  International Physical Activity questionnaire score
fear for hypoglycaemia | between 36.0-38.6 weeks
  the Hypoglycaemia Fear Survey II
fear for hyperglycaemia | between 36.0-38.6 weeks
  self-designed questionnaire on fear for hyperglycaemia
symptoms of depression | baseline, between 36.0-38.6 weeks and 6-24 weeks postpartum
  the 20-item Center for Epidemiologic Studies-Depression (CES-D) , questionnaire, max. score 60 (the higher the more symptoms of depression)
symptoms of anxiety | baseline, between 36.0-38.6 weeks and 6-24 weeks postpartum
  validated six-item short-form STAI questionnaire on anxiety, max. score of 24 (the higher the more anxiety)
user-friendliness of CGM | between 36.0-38.6 weeks
  self-designed questionnaire on the user-friendliness of continuous glucose monitoring (CGM)
user-friendliness of CGM compared to oral glucose tolerance test (OGTT) | between 6-24 weeks postpartum
  self-designed questionnaire on the user-friendliness of continuous glucose monitoring (CGM) compared to OGTT
duration of breastfeeding | postpartum between 6-24 weeks
  breastfeeding duration (exclusive or half formula) duration in months
rate of hypercholesterolemia | postpartum between 6-24 weeks
  lipid profile with LDL-cholesterol and Triglycerides
night glucose time in range between 70-180mg/dl | postpartum between 6-24 weeks
  glucose time in range between 70-180mg/dl from 00 til 6am
day glucose time in range between 70-180mg/dl | postpartum between 6-24 weeks
  glucose time in range between 70-180mg/dl from 6am till 00
day glucose time in range <70mg/dl | postpartum between 6-24 weeks
  glucose time below 70-mg/dl from 6am till 00
night glucose time in range <70mg/dl | postpartum between 6-24 weeks
  glucose time below 70-mg/dl from 00 till 6am
night glucose time in range >180mg/dl | postpartum between 6-24 weeks
  glucose time above 180mg/dl from 00 till 6am
day glucose time in range >180mg/dl | postpartum between 6-24 weeks
  glucose time above 180mg/dl from 6am till 00

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (14):
  - OLV Aalst-Asse, Aalst, Oost-Vlaanderen
  - UZA, Antwerp
  - ZNA Antwerpen, Antwerp
  - Imelda Bonheiden, Bonheiden
  - AZ St Jan Brugge, Bruges
  - Erasme, Brussels
  - UZ Gent, Ghent
  - AZ St Lucas Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - AZ St Maarten Mechelen, Mechelen
  - AZ Oostende, Ostend
  - Vitaz, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No